CLINICAL TRIAL: NCT06715241
Title: A MULTICENTER, SEEKING SIGNAL, RANDOMISED, OPEN-LABEL PHASE II OF RELATLIMAB AND NIVOLUMAB VS NIVOLUMAB ALONE IN LOCALLY ADVANCED CERVICAL CANCERS
Acronym: COLIBRI-2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GINECO-CE111b; 2024-514032-25-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: LOCALLY ADVANCED CERVICAL CANCERS
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Nivolumab and relatlimab (Experimental)
  Interventions: Combination Product: combination of relatlimab and nivolumab wich are two immunotherapy treatments
- Arm B: Nivolumab only (Other)
  Interventions: Other: Nivolumab alone

INTERVENTIONS:
Combination Product: combination of relatlimab and nivolumab wich are two immunotherapy treatments — Induction: Nivolumab 360 mg/relatlimab 360 mg fixed dose combination, IV, 6 weeks Off treatment period: 4 to 6 weeks Maintenance: Nivolumab 480 mg/relatlimab 480 mg fixed dose combination, IV 13 cycles (Q4W): 52 weeks
  Arms: Arm A: Nivolumab and relatlimab
Other: Nivolumab alone — Induction: Nivolumab alone 360 mg, IV2 cycles (Q3W): 6 weeks Off treatment period: 4 to 6 weeks Maintenance: Nivolumab alone 480 mg, IV, 13 cycles (Q4W): 52 weeks
  Arms: Arm B: Nivolumab only

SUMMARY:
Multicenter, open-label, randomized, seeking signal (non-comparative), Phase II aiming to assess the clinical activity of the combination relatlimab + nivolumab in locally advanced cervical cancer eligible to standard CCRT

DETAILED DESCRIPTION:
Primary Objective

* To evaluate the clinical activity of relatlimab and nivolumab induction treatment before standard CCRT in locally advanced cervical cancer

Secondary Objectives

* To further document the clinical activity of relatlimab and nivolumab
* To document the safety of the proposed combination in the target population

Exploratory Objectives

* To identify candidate biomarkers that may correlate with likelihood of clinical benefit/response using serial blood and tumor sample collection.
* To explore the factors (including biomarkers) that may influence response (where response is defined broadly to comprise efficacy, tolerability or safety) or to explore mechanisms of resistance to study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥18 years at time of inform consent signature.
* Patients must have histologically confirmed diagnosis of cervical squamous or adenosquamous carcinoma stage IIB to IVA according to FIGO 2018 (Appendix 1) and no evidence of metastatic disease (M0). Note: Nodal staging may be either surgical or by imaging (MRI/PET-CT) with pathological lymph node size defined by a short-axis diameter of ≥10mm (axial plane) or FDG uptake greater than that of the surrounding tissue and corresponding to the LN structure on CT when CT was performed for PETCT analysis.
* Patients must be naïve from prior anti-cancer treatment (all type) and eligible to standard CCRT as per standard practice and investigator' judgement.
* Known HPV status as per local assessment.
* Patient accepting to undergo a new cervix biopsy and with at least one lesion with a diameter ≥10 mm, visible by medical imaging and accessible to percutaneous sampling (needle biopsies 16 gauge or larger) that permit core needle biopsy (ideally 4 cores) without unacceptable risk of a major procedural complication.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Appendix 2).
* Adequate organ and marrow function with following lab values within 7 days before C1D1:

  * Absolute neutrophil count (ANC) ≥1500/μL
  * White blood cell (WBC) >3000/μL
  * Platelets ≥100 000/μL
  * Hemoglobin (Hb) ≥9 g/dL
  * Total bilirubin ≤1.5× upper limit of normal (ULN) unless due to Gilbert's syndrome
  * ASAT /ALAT ≤3 ULN
  * Creatinine ≤1.5 within normal limit, or
  * Creatinine clearance ≥ 40 mL/min according to CKD-EPI formula (Appendix 3)
  * Troponin T or I < 2 x ULN
* Adequate cardiovascular function documented by:

  * QTc interval <450 msec.
  * Left ventricular Ejection fraction > 50% based on screening echocardiogram (ECHO) or multigated acquisition scan (MUGA).
  * Controlled blood pressure (BP, <150/90mmHg), with or without current antihypertensive treatment.
  * No congestive heart failure New York Heart Association class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias (eg, ventricular flutter, ventricular fibrillation, Torsades de pointes).
  * No stroke (including transient ischemic attack [TIA]), myocardial infarction, or other clinically significant ischemic event within 12 months before first dose.
  * No prior history of myocarditis.
* Women of childbearing potential

  * must have a negative serum pregnancy test within 7 days prior C1D1 and use adequate contraceptive methods (for example, intrauterine device [IUD], birth control pills unless clinically contraindicated, or barrier device - see Appendix 4) beginning 2 weeks before the first dose of study drugs and for up to 6 months after the final dose of study drugs (i.e., 30 days [duration of ovulatory cycle] plus the time required for relatlimab and nivolumab to undergo approximately five halflives).
  * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries, fallopian tubes, and/or uterus).
* Ability to understand and sign informed consent and willingness to comply with the study procedures before study entry.
* Covered by a medical insurance.

Exclusion Criteria:

* Evidence or treatment for another malignancy within 3 years prior to study entry. Curatively treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia is allowed.
* History of severe allergic or other hypersensitivity reactions to:

  * chimeric or humanized antibodies or fusion proteins,
  * biopharmaceuticals produced in Chinese hamster ovary cells, or
  * any component of the study treatments formulation.
* Patients with:

  * Active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) unless their HBV is stably controlled on nucleoside analogs (eg entecavir or tenofovir) which will be continued for the duration of the study. Note: Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. HBV DNA test must be performed in these patients prior to C1D1.
  * Active hepatitis C. Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA, or
  * HIV infection. Patients with prior organ or bone marrow transplant.
* Patients with active, suspected or history of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis (see Appendix 5 for a more comprehensive list of pre-existing autoimmune diseases and immune deficiencies) with the following exceptions:

  * patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone,
  * patients with controlled Type 1 diabetes mellitus,
  * patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    * rash must cover less than 10% of body surface area (BSA).
    * disease is well controlled at baseline and only requiring low potency topical steroids.
    * no acute exacerbations of underlying condition within the previous 12 months requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency or oral steroids.
* Patients not respecting the minimal washout period or anticipation of need during the study of the following medications:

  1. For "Systemic immunosuppressive medication (e.g.corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents)", a minimal wash out period before C1D1 ≥ 2 weeks is requested.

     But use during the study is not allowed with the exceptions of intranasal, inhaled, or topical corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10mg/day of prednisone, or an equivalent corticosteroid.
  2. For "Systemic immunostimulatory (e.g., interferons and IL-2), a minimal wash out period ≥ 4 weeks or 5 * t(1/2) of medication whichever is longer.

But use during the study is not allowed.

* Patients with any serious or uncontrolled medical disorder that, in the opinion of the investigator, may have increased the risk associated with trial participation or trial treatment administration, impaired the ability of the patients to receive protocol therapy, or interfered with the interpretation of trial results.
* Patients have received a live/attenuated vaccine within 30 days of C1D1 (inactivated vaccines were permitted).
* Pregnant or lactating women.
* Patients deprived of liberty, under guardianship, or under curatorship.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2024-12-11 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | From the date of randomization until patients operated with late complete debulking surgery, assessed up 100 days
  Objective response rate at the end of the 6-week induction period is defined as the rate of patients with CR or PR as per RECIST V1.1 at the end of the induction period.
  Response will be assessed according to RECIST v1.1 criteria as per investigator assessment.
  ORR-6w will be derived as a binary variable (success/failure), based on the following rules:
  * Patients showing an objective response based on RECIST tumoral evaluation performed at the end of the induction period will be considered in " success ".
  * Patients showing a progressive disease based on RECIST tumoral evaluation performed at the end of the induction period will be considered in " failure ".
  * Patients with no tumoral evaluation at the end of the induction period and with early death or clinical progression or treatment discontinuation due to toxicity will be considered in " failure ".
  * Patients who do not meet any of the conditions above will be consider as " non evaluable " for the primary endpoint.

SECONDARY OUTCOMES:
Progression Free survival (PFS) | From the date of randomization until patients operated with late complete debulking surgery, assessed up 100 days
  PFS is defined as the time from randomization until the date of event defined as the first objective documented progression, according to investigator assessment of RECIST v1.1 or death (by any cause in the absence of progression). Patients who have not progressed or died at the time of analysis will be censored at the time of the latest date of assessment from their last evaluable RECIST assessment.
Time to local progression (TTlP) | From the date of randomization until patients operated with late complete debulking surgery, assessed up 100 days
  TTlP will be measured from the date of randomization to the date of event defined as the 1st local progression, and censored at the date of last tumor assessment for patients without event at the time of the analysis.
Time to metastatic progression (TTmP) | From the date of randomization until patients operated with late complete debulking surgery, assessed up 100 days
  TTmP will be measured from the date of randomization to the date of event defined as the 1st metastatic progression, and censored at the date of last tumor assessment for patients without event at the time of the analysis. Patients with no post-baseline tumoral evaluation (e.g withdrawal of consent) will be censored at day 1 for the evaluation of PFS, TTlP and TTmP.
Overall Survival (OS) | From the date of randomization until patients operated with late complete debulking surgery, assessed up 100 days
  OS isis defined as the time from the date of randomization until death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.
ORR after CCRT/at the end of the maintenance period | From the date of randomization until patients operated with late complete debulking surgery, assessed up 100 days
  It is defined as the rate of patients with CR or PR as per RECIST V1.1 after CCRT/at the end of the maintenance period. ORR after CCRT/ at the end of the maintenance period will be derived in the same way as ORR-6w.

CONTACTS AND LOCATIONS:
Locations (30):
- France (30):
  - ICO Paul Papin, Angers
  - Sainte-Catherine Institut du Cancer Avignon-Provence, Avignon
  - CHRU Besançon - Hôpital Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - CHU de BREST - Hôpital Cavale Blanche, Brest
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - CHU de Dijon, Dijon
  - Soumya.Anane@chicreteil.fr, Dijon
  - CHRU Lille - Hôpital Jeanne de Flandre, Lille
  - Centre Oscar Lambret, Lille
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Groupe Hospitalier Diaconesses - Croix Saint-Simon, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre CARIO - HPCA, Plérin
  - CHU de Poitiers - Hôpital de la Milétrie, Poitiers
  - Centre Eugène Marquis, Rennes
  - CHU Saint-Etienne - Pôle de Cancérologie, Saint-Etienne
  - ICO - Centre René Gauducheau, Saint-Herblain
  - ICANS - Institut de cancérologie Strasbourg Europe, Strasbourg
  - CHU STRASBOURG - Hôpital de Hautepierre, Strasbourg
  - Oncopole Claudius Regaud, Toulouse
  - Recherche Oncologique Clinique 37 (ROC 37), Tours
  - ICL - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif